CLINICAL TRIAL: NCT06847906
Title: Evaluating the Reach of Clinical Decision Support for Patients With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (AHA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-1154; 23SCISA1144584 (Other: American Heart Association)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Decision Support Systems, Clinical; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Compare two different types of a virtual CDS tool in a randomized pilot study at one health system.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iteratively designed (new) clinical decision support tool for virtual visits (Experimental)
  Interventions: Other: Iteratively designed (new) clinical decision support tool for virtual visits
- Traditional clinical decision support tool (Experimental)
  Interventions: Other: Traditional clinical decision support tool

INTERVENTIONS:
Other: Iteratively designed (new) clinical decision support tool for virtual visits — The new, iteratively designed clinical decision support tool includes the traditional CDS along with links to supportive tipsheets, which include one for providers on how to add an order for patients to upload vitals in their electronic health record, and one that walks patients through how to upload vitals on their own.
  Arms: Iteratively designed (new) clinical decision support tool for virtual visits
Other: Traditional clinical decision support tool — The traditional CDS tool is the usual care intervention, and does not include links to tipsheets to support virtual patient care.
  Arms: Traditional clinical decision support tool

SUMMARY:
To work best, clinical decision support tools (CDS) must be timed to provide support when healthcare decisions are made, which includes virtual visits (phone or video). Unfortunately, most CDS tools are either missing from virtual visits or not designed for the unique context of virtual visits (e.g., availability of physical assessments and labs, different workflows), which could generate new inequities for patients more likely to use virtual visits. The objective of this study is to test the reach, feasibility and acceptability of a new CDS tool for heart failure with reduced ejection fraction (HFrEF) during virtual visits. This new CDS tool was developed through an iterative design process, and will be compared to an existing HFrEF CDS tool in a randomized pilot study at outpatient cardiology clinics throughout the UCHealth system.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects are potential users of the CDS, specifically clinicians with prescribing privileges who practice at one of the health system's (UCHealth) outpatient cardiology clinics. Because we are observing their prescribing behaviors in a virtual care setting (phone or video), we are also evaluating patient characteristics which could influence their prescribing decisions.

Exclusion Criteria:

* Clinicians who do not practice in a UCHealth cardiology clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of CDS alerts resulting in the prescription of a recommended medication | 6 months
  The primary outcome is number of CDS alerts that resulted in the prescription of the medication recommended by the CDS alert. Recommended medications include either evidence-based beta blockers, sacubitril/valsartan, mineralocorticoid receptor antagonists or sodium/glucose cotransport 2 inhibitors. Prescriptions will be based on actual prescription orders instead of clinician-stated responses, given the latter may overestimate effectiveness.

SECONDARY OUTCOMES:
Number of patients the CDS alerted for | 6 months
  This outcome evaluates the reach of the CDS by counting the number of patients that the CDS alerted for.
Number of times a prescriber ordered at-home vitals | 6 months
  This outcome will count the number of times a prescriber orders patients to take their vitals at home after being exposed to the CDS tool.
Number of patients who upload their vitals in the patient portal | 9 months
  This outcome will count the number of patients who upload their vitals into the electronic medical record.
Number of alerts that were not outright dismissed | 6 months
  This outcome will help investigators understand if the CDS id being used or dismissed.
Number of prescription orders for guideline directed medical therapy (GDMT) for heart failure | 6 months
  This outcome measures the number of prescriptions for each of the four categories of GDMT: evidence-based beta blockers, sacubitril/valsartan, mineralocorticoid receptor antagonists or sodium/glucose cotransport 2 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Trinkley, PharmD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth Primary Care and Cardiology Outpatient Clinics, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.